CLINICAL TRIAL: NCT04403399
Title: Cholinergic Mechanisms of Gait Dysfunction in Parkinson's Disease Experiment 3 - Project #3
Brief Title: Crossover Target Engagement Study of Cholinergic Mechanisms of Gait Dysfunction in Parkinson's Disease (Project #3 - Experiment 3 [UdallP3E3])
Acronym: UdallP3E3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Roger L. Albin, Professor of Neurology, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00093188-a
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Varenicline then Placebo (Experimental): Varenicline 0.5 mg BID orally for 3 weeks, followed by a 3-week washout period, then placebo BID orally for 3 weeks
  Interventions: Drug: Varenicline; Drug: Placebo
- Placebo then Varenicline (Experimental): Placebo BID orally for 3 weeks, followed by a 3-week washout period, then Varenicline 0.5 mg BID orally for 3 weeks
  Interventions: Drug: Varenicline; Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Initial 0.25 mg oral dose of varenicline administered with monitoring over 4 hours, then total daily dose escalated over the next 2 days until final 0.5 mg BID oral varenicline administered for the remaining 3 weeks.
  Other Names: Chantix
Drug: Placebo — Initial placebo oral dose administered with monitoring over 4 hours, then total daily dose escalated over the next 2 days until final placebo BID dosing administered orally for the remaining 3 weeks.

SUMMARY:
With an appropriate oral dose of Varenicline (VCN) identified from experiments 1 & 2 of the study (see NCT02933372), the investigators will administer VCN to Parkinson Disease (PD) participants to determine if VCN improves walking speed and measures of balance. PD participants will receive VCN or a placebo (fake drug) for 3 weeks to assess the effects of VCN administration on gait speed and balance. Participants will undergo examinations to assess the intensity of their Parkinsonism and asked questions to assess their mood and thinking.

DETAILED DESCRIPTION:
To demonstrate that α4β2* nAChRs are appropriate therapeutic targets in Parkinson's Disease (PD), it is necessary to study key pharmacokinetic-pharmacodynamic features of α4β2* nAChR in the context of the PD brain with loss of nerve cells that produce the neurotransmitter acetylcholine, a pathologic environment in which they may exhibit unique features. This personalized medicine approach focuses our studies on the subgroup of PD subjects with loss of nerve cells that produce the neurotransmitter acetylcholine identified by Project II and the Clinical Resource Core. The investigators will assess α4β2* nAChR features using PET imaging with the α4β2* nAChR ligand [18-Fluorine]flubatine, subacute administration of the α4β2* nAChR partial agonist Varenicline (VCN), and laboratory measures of gait, balance, and attention. The investigators will use [18-Fluorine] flubatine PET to assess VCN occupancy of brain α4β2* nAChRs (experiments 1 & 2). VCN will be administered to both PD participants (experiment 1) and healthy controls (experiment 2) and both populations will undergo a flubatine PET scan to assess VCN occupancy. Using this PET data to select an appropriate VCN dose, the investigators will perform a pharmacodynamic study (experiment 3) with subacute VCN administration to determine if α4β2* nAChR stimulation improves laboratory measures of gait function, postural control, and attentional function in PD subjects with loss of nerve cells that produce the neurotransmitter acetylcholine.

ELIGIBILITY:
Inclusion Criteria:

1. PD diagnosis will be based on the United Kingdom Parkinson's Disease Society Brain Bank Research Center (UKPDSBRC) clinical diagnostic criteria. The investigators will enrich the cohort by recruiting subjects at modified Hoehn and Yahr stages 2 or higher, duration of motor disease 5 years or longer, age >65 years, or the Postural Instability and Gait Disorder (PIGD) phenotype. Duration of motor disease will be defined as the time between onset of motor symptoms and time of entry into the study. The PIGD phenotype is defined as described previously. PD subjects with defined cholinergic deficits will be recruited as described in Project II. PD subjects will have cortical cholinergic deficits based on 5th percentile cutoff of the normal controls as defined previously.
2. Stable dopaminergic replacement therapy for 3 months prior to enrollment and expected to maintain stable dopaminergic therapy for duration of study participation.

Exclusion Criteria:

1. Other disorders which may resemble PD with or without dementia, such as vascular dementia, normal pressure hydrocephalus, progressive supranuclear palsy, multiple system atrophy, corticobasal ganglionic degeneration, or toxic causes of parkinsonism. Prototypical cases have distinctive clinical profiles, like vertical supranuclear gaze palsy, early and severe dysautonomia or appendicular apraxia, which may differentiate them from idiopathic PD. The use of the UKPDSBRC clinical diagnostic criteria for PD will mitigate the inclusion of subjects with atypical parkinsonism and all participants will undergo [11-Carbon]dihydrotetrabenazine PET to confirm striatal dopaminergic denervation.
2. Subjects on neuroleptic, anticholinergic (trihexphenidyl, benztropine), or cholinesterase inhibitor drugs.
3. Current or previous (within last 6 months) use of any product or medication containing nicotinic agents,including use of tobacco products such as cigarettes, cigars, pipes, chewing tobacco, etc., electronic cigarettes, over-the-counter nicotine patches, chewing gum containing nicotine, or varenicline.
4. Evidence of a stroke or mass lesion on structural brain imaging (MRI).
5. Participants in whom magnetic resonance imaging (MRI) is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant.
6. Severe claustrophobia precluding MR or PET imaging
7. Subjects limited by participation in research procedures involving ionizing radiation.
8. Pregnancy (test within 48 hours of each PET session) or breastfeeding.
9. Significant risk of cardiovascular event.
10. Active, significant mood disorder.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger L Albin, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mancini M, Carlson-Kuhta P, Zampieri C, Nutt JG, Chiari L, Horak FB. Postural sway as a marker of progression in Parkinson's disease: a pilot longitudinal study. Gait Posture. 2012 Jul;36(3):471-6. doi: 10.1016/j.gaitpost.2012.04.010. Epub 2012 Jun 29. PMID 22750016

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline Then Placebo: Patients will take varenicline initially for 3 weeks, then after a 3 week washout period, they will switch to placebo for 3 weeks.
- Placebo Then Varenicline: Patients will take placebo initially for 3 weeks, then after a 3 week washout period they will switch to varenicline for 3 weeks.
Period: Period 1
Arm/Group | Varenicline Then Placebo | Placebo Then Varenicline
Started | 18 | 16
Completed | 18 | 16
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Varenicline Then Placebo | Placebo Then Varenicline
Started | 18 | 16
Completed | 18 | 15
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Then Varenicline: Patients will take placebo initially for 3 weeks, then after a 3 week washout period, they will switch to varenicline for 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Varenicline Then Placebo | Placebo Then Varenicline | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (5.7) | 64.2 (5.3) | 66.3 (5.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 15 | 13 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 17 | 16 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 16 | 34
Age at Diagnosis of Parkinson's Disease [Mean (Standard Deviation); unit: years] | 61.3 (6.66) | 57.7 (7.22) | 59.6 (7.06)
MDS-UPDRS III [Mean (Standard Deviation); unit: units on a scale] — Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III (motor examination) includes 18 items (33 scores). Each item scores from 0 (normal) to 4 (severe) and total score is obtained from the sum of the corresponding item scores. The minimum is 0, maximum is 132, with higher scores indicating more disability.
  units on a scale | 33.2 (13.92) | 30.7 (12.4) | 32.0 (13.07)
Geriatric Depression Scale [Mean (Standard Deviation); unit: units on a scale] — Geriatric Depression Scale (GDS) is a 30-item questionnaire (long form) to measure depression in the older population. Participants are asked to respond yes or no to how they felt over the past week. Scores range from 0 to 30, with higher scores indicating more severe depression.
  units on a scale | 2.4 (2.06) | 4.3 (4.19) | 3.3 (3.34)
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — Montreal Cognitive Assessment (MoCA) is a questionnaire assessing cognitive dysfunction. It assesses attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The score ranges from 0 to 30, with higher scores indicating more severe cognitive impairment.
  units on a scale | 27.2 (2.37) | 26.8 (1.97) | 27.0 (2.17)

OUTCOME MEASURES:

1. Primary Outcome: Gait Speed
Description: Gait speed, how fast a person can walk down a corridor, at normal pace with no distractors (i.e., no dual task).
Time Frame: end of each period: 22 and 64 days
Population: All randomized participants were included in the mixed effects model. One participant randomized to the placebo then varenicline group was withdrawn by the physician early in period 2; 1 participant randomized to the varenicline then placebo group did not complete the gait assessment in period 2.
Measure: Least Squares Mean (Standard Error); unit: cm/s
Groups:
- Varenicline: 0.5 mg PO BID varenicline for 3 weeks (beginning with a 0.25 mg dose and escalated over the next 2 days)
- Placebo: placebo given PO BID for 3 weeks
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 33 | 33
cm/s | 121.27 (1.36) | 124.89 (1.36)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -3.62

2. Primary Outcome: JERK
Description: JERK is the time based derivative of spontaneous lower trunk accelerations during standing. It was assessed with the Ambulatory Parkinson's Disease Monitoring (APDM) wearable sensor system (APDM Wearable Technologies, Inc.) using the iSWAY protocol, with participants standing on a foam pad with eyes closed. JERK was calculated using the manufacturer's software (Mobility Lab Version 1).
Time Frame: end of each period: 22 and 64 days
Population: All randomized participants were included in the mixed effects model. One participant randomized to the placebo then varenicline group was withdrawn by the physician early in period 2; two participants randomized to the varenicline then placebo group did not complete the iSWAY protocol in period 2.
Measure: Least Squares Mean (Standard Error); unit: m^2/sec^5
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 33 | 32
m^2/sec^5 | 0.97 (0.20) | 1.04 (0.20)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority; p = 0.73, Mixed Models Analysis; Mean Difference (Final Values) = -0.07

3. Secondary Outcome: Attention
Description: Attention function will be measured with a standard computer test, the Sustained Attention Test (SAT), without a distractor condition. Results are reported as the vigilance index, a measure that corrects estimates of accurate detection with penalties for false detection and not confounded by errors of omission. (Frey PW, Colliver JA. Sensitivity and responsivity measures for discrimination learning. Learn Motiv 1973; 4:327-342.) The minimum score is -1.00 (indicating that all recorded responses were misses or false alarms) and maximum is +1 (indicating that all recorded responses were hits or correct rejections). Higher values indicate better attentional performance.
Time Frame: end of period: days 22 and 64
Population: All randomized participants with at least one post-treatment value were included in the mixed effects model. Six participants (1 in the placebo then varenicline, 6 in the varenicline then placebo) were unable to pass practice trials due to delayed response time (task not completed at all visits). Technical errors resulted in missing data for 2 placebo and 1 varenicline participants; 3 varenicline participants requested skipping task due to physical ailments.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 23 | 26
units on a scale | 0.73 (0.06) | 0.66 (0.06)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Final Values) = 0.08

ADVERSE EVENTS:
Time Frame: 9 weeks (3 weeks in period 1, 3 weeks in washout, 3 weeks in period 2)
Arm/Group | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/34 | 1/34
Other Adverse Events (participants affected / at risk) | 17/34 | 8/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=34) | Placebo (N=34)
Syncope, unspecified (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitus (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=34) | Placebo (N=34)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 1 (1)
Lightheadedness (Nervous system disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Cramping in left leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Decreased reflexes in distal lower extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1)
Difficulty walking (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foggy/Forgetfulness (Nervous system disorders) | 1 (1) | 1 (1)
Hammer toes (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Inability to sleep (Psychiatric disorders) | 1 (1) | 0 (0)
Increase in appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increase in PD medication "off" time (Nervous system disorders) | 3 (3) | 0 (0)
Increase stiffness in hands (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Increased tremors (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Involuntary movements (Nervous system disorders) | 1 (1) | 0 (0)
Pain in shoulder, pelvic (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
New onset of perception difficulty (Nervous system disorders) | 1 (1) | 0 (0)
Tendon tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ringing in ears (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Systolic ejection murmur (Cardiac disorders) | 1 (1) | 0 (0)
Tiredness (General disorders) | 1 (1) | 1 (1)
Toothache (General disorders) | 1 (1) | 0 (0)
Vasovagal syncope (Nervous system disorders) | 1 (1) | 0 (0)
Vivid dreams (Psychiatric disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT04403399/SAP_000.pdf
  • Study Protocol (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT04403399/Prot_001.pdf